CLINICAL TRIAL: NCT01105949
Title: An Evaluation of Two Novel Breathe Right Nasal Strip Prototypes on Nasal Patency
Brief Title: An Evaluation of Two Novel Nasal Strip Prototypes on Nasal Patency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3560645
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Volunteer
Keywords: nasal patency; acoustic rhinometry; nasal strip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Marketed nasal strip (Other): Marketed nasal strip
  Interventions: Device: Marketed nasal strip
- NexGen JB Organic PET/PE (Experimental): NexGen JB Organic PET/PE, prototype nasal dilator strip
  Interventions: Device: NexGen JB Organic PET/PE
- NexGen AB 2R11 (Experimental): NexGen AB 2R11
  Interventions: Device: NexGen AB 2R11

INTERVENTIONS:
Device: Marketed nasal strip — Marketed nasal strip
  Arms: Marketed nasal strip
Device: NexGen AB 2R11 — Nasal strip prototype
  Arms: NexGen AB 2R11
Device: NexGen JB Organic PET/PE — Nasal strip
  Arms: NexGen JB Organic PET/PE

SUMMARY:
The results of this study will help in the development of a new type of nasal strip for management of nasal congestion and snoring.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history

Exclusion Criteria:

* Currently experiencing cold or flu
* History of perennial or allergic rhinitis or rhinitis medicamentosa
* Evidence of nasal polyps as documented by anterior rhinoscopy
* Evidence of significant nasal tract structural malformations including a severe deviated septum (where subjects are indicated for surgery) or a concha bullosa as documented by anterior rhinoscopy
* Visible open sores, sunburn, irritation, eczema or chronic skin condition on the face to nose
* Bacterial sinusitis infection during 2 weeks prior to entry in the baseline phase of the study
* Any other condition that in the opinion of the investigator would have an affect on nasal breathing
* Use of any product containing menthol within two hours prior to any subjective measures involved in the study
* Had an allergic contact dermatitis on the face within 30 days prior to entry
* History of chronic or active skin or other immunologic (rheumatoid, psoriasis) disease
* History of skin cancer
* Use of antibiotics or alpha adrenergic drugs (all forms) within 1 week prior to entry in the baseine phase of the study
* Use of glucocorticosteroids (all forms) within 1 month prior to entry in the baseline phase of the study
* Any current treatment which in the opinion of the investigator will affect nasal congestion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in minimum cross sectional area (second restriction) of the nasal valve using acoustic rhinometry | baseline to within 2 hours post application
Change from baseline in total nasal volume of the nose using acoustic rhinometry | baseline to within 2 hours post application

SECONDARY OUTCOMES:
Nasal airway breathing as measured by Posterior Rhinomanometry | Baseline to 2 hours
Nasal airway breathing as measured by Peak Nasal Inspiratory Flow (PNIF) | Baseline to 2 hours
Subjective perceptions of airway breathing | Baseline to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Common Cold Centre, Cardiff, Wales, United Kingdom

REFERENCES:
- [Derived] Ward J, Ciesla R, Becker W, Shanga GM. Randomized Trials of Nasal Patency and Dermal Tolerability With External Nasal Dilators in Healthy Volunteers. Allergy Rhinol (Providence). 2018 Oct 5;9:2152656718796740. doi: 10.1177/2152656718796740. eCollection 2018 Jan-Dec. PMID 30305980